CLINICAL TRIAL: NCT01869868
Title: Neurobiological Changes and Clinical Outcome When Treating Depression With Electroconvulsive Therapy.
Brief Title: Neurobiological Changes When Treating Depression With Electroconvulsive Therapy - a Longitudinal Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Pia Nordanskog, MD, Linkoeping University
Other Study IDs: LIU2012/310-31; LinkoepingUniversity (Other: LinkoepingUniversity)
Record Dates: First submitted 2013-06-02; First posted 2013-06-05 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Depression, ECT

SUMMARY:
The purpose of this study is to determine functional and structural changes in brain following treatment of severe depression with electroconvulsive therapy with correlation to clinical outcome. Our hypothesis is that there are state-dependent changes in functional connectivity within specific neurocircuits systems, as well as structural plasticity changes in hippocampus, when recovering from depression.

DETAILED DESCRIPTION:
The study is a prospective, within-subject, observational follow-up study in individuals with depression who receive electroconvulsive therapy (ECT)at a psychiatric clinic. We will use a consecutive sampling method and patient referred for ECT by their psychiatrist will be screened for inclusion and asked for participation. Both in - and outpatients can be included. At three occasions (before treatment, after four week and after three months) patients will be assessed with clinical ratings, cognitive tests, functional and structural magnetic resonance imaging and biomarkers for cell proliferation.

ELIGIBILITY:
Inclusion Criteria:

* major depressive disorder
* depressive episode in bipolar disorder
* age 18 - 65 years

Exclusion Criteria:

* alcohol- and/or drug dependence or abuse in the past 3 months
* severe/life-threatening medical disease
* pregnancy
* type I diabetes
* neurodegenerative disorder
* inability to give written informed consent to participation in the study
* contradiction to MRI scanning.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with depression referred for ECT.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Measures of hippocampal volume assessed by structural MRI | Three months
fMRI BOLD resting state functional connectivity | 3 month
fMRI BOLD responses during execution of emotional and reward processing tasks | 3 months
Biomarkers of cell proliferation | 3 months

SECONDARY OUTCOMES:
Relation between neurobiological changes and clinical and cognitive outcome | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Linkoeping University, Linkoeping University Hospital, Linköping, Östergötland County, Sweden